CLINICAL TRIAL: NCT00268905
Title: A Phase Ib Open-Label, Two-Arm, Dose-Finding Study of E7389 in Combination With Carboplatin in Patients With Solid Tumors
Brief Title: A Dose-Finding Study of E7389 in Combination With Carboplatin in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7389-A001-104
Record Dates: First submitted 2005-12-21; First posted 2005-12-23 (Estimated); Results first posted 2013-01-25 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — eribulin

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: E7389 + carboplatin AUC 5
- 2 (Experimental)
  Interventions: Drug: E7389 + carboplatin AUC 6
- 3 (Experimental)
  Interventions: Drug: E7389+carboplatin AUC 6

INTERVENTIONS:
Drug: E7389 + carboplatin AUC 5 — Patients will receive E7389 before (Schedule A) or after (Schedule B) carboplatin AUC 5 infusion. E7389 will be administered as a 2-5 minute intravenous (IV) bolus infusion at a starting dose of 0.7 mg/m^2 on Days 1 and 8 every 21 days. Carboplatin 5 AUC will be administered as a 30-minute IV infusion on Day 1 every 21 days. Dose escalation will be performed in cohorts of three patients per dose level per schedule.
  Arms: 1
Drug: E7389 + carboplatin AUC 6 — After MTD is reached with carboplatin AUC 5, dose escalation of E7389 in combination with carboplatin at AUC 6 will begin at one dose level below MTD, using the preferred schedule (A or B).
  If carboplatin AUC 6 with E7389 is tolerated, the MTD reached will be used to enroll 20 additional patients with Stage IIIB or IV non-small cell lung cancer (NSCLC). If carboplatin AUC 6 is not tolerated, these patients will be enrolled at the MTD determined with the combination of E7389 and carboplatin AUC 5.
  Arms: 2
Drug: E7389+carboplatin AUC 6 — In a population of patients who had generally received multiple prior chemotherapies, the eribulin MTD has been determined to be 1.1 mg/m2 in combination with carboplatin at an AUC of 6. The first-line NSCLC patients in the extension arm may tolerate a higher dose of eribulin, because they have not been exposed to the toxicity of other chemotherapies. To investigate this possibility, the dose of eribulin will be increased to 1.4 mg/m2 for subsequent patients, if the first six of these patients do not experience a DLT during their first cycle of eribulin at 1.1 mg/m2 and carboplatin at AUC 6 combination therapy. If no more than one of the first six patients experience a DLT during the first cycle with the 1.4 mg/m2 dose of eribulin, then the 1.4 mg/m2 dose will be considered the recommended dose for front-line NSCLC therapy and the remaining patients will be treated using this dose.
  Arms: 3

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD) and to explore the safety and anti-tumor activity of E7389 in combination with carboplatin in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a Phase Ib open-label, two-arm, dose-finding study of E7389 in combination with carboplatin in patients with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years of age.
2. Patients with an Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1.
3. Patients with a life expectancy of ≥ three months.
4. Patients with adequate renal function as evidenced by serum creatinine ≤ 2.0 mg/dL or calculated creatinine clearance ≥ 40 mL/min per the Cockcroft and Gault formula.
5. Patients with adequate bone marrow function as evidenced by absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L, hemoglobin ≥ 10.0 g/dL (this may have been corrected by transfusion or growth factors) and platelet count ≥ 100 × 10^9/L.
6. Patients with adequate liver function as evidenced by bilirubin ≤ 1.5 mg/dL and alkaline phosphatase (ALP), alanine transaminase (ALT) and aspartate aminotransferase (AST) ≤ 3 times the upper limits of normal (ULN) (in the case of liver metastases ≤ 5 x ULN), unless there are bone metastases, in which case liver specific alkaline phosphatase must be separated from the total and used to assess the liver function instead of the total alkaline phosphatase. to assess the liver function instead of the total alkaline phosphatase.
7. Patients willing and able to comply with the study protocol for the duration of the study.
8. Written informed consent prior to any study-specific screening procedures with the understanding that the patient may withdraw consent at any time without prejudice.

For patients in the dose finding phase, the following additional inclusion criteria must be fulfilled:

1. Patients with pathologically diagnosed, histologically or cytologically confirmed advanced solid tumor, that has progressed following standard therapy or for which no standard therapy exists (including surgery or radiation therapy).
2. Patients with disease progression despite standard therapy or have disease for which no standard therapy exists.
3. Patients with ≤ Grade 2 chemotherapy or radiation-related toxicities except alopecia.

For NSCLC patients at the MTD, the following additional inclusion criteria must be fulfilled:

1. Patients with pathologically diagnosed, histologically or cytologically confirmed advanced NSCLC (Stage IIIB or IV) with measurable disease, not amenable to surgical or radiation treatment.
2. Patients with no prior chemotherapy for NSCLC including neoadjuvant or adjuvant treatment.

Exclusion Criteria:

1. Patients are excluded if they have received any of the following within three weeks prior to first study treatment: investigational drugs, immunotherapy, gene therapy, hormone therapy (except leuprolide, and megestrol acetate for appetite stimulation), other biological therapy, chemotherapy or radiation. Patients with major surgery without full recovery or major surgery within 3 weeks prior to first study treatment are also excluded. Patients must have recovered from any previous major therapy-related toxicity (Grade 3 or 4) to < Grade 2 at study entry (except for neuropathy).
2. Patients who have received radiation ≤ 3 weeks prior to study enrollment, whose marrow exposure has exceeded 30% or who have not recovered from the toxic effects of the treatment prior to study enrollment (except for alopecia).
3. Patients who have received prior high dose chemotherapy with hematopoietic stem cell rescue or stem cell or bone marrow transplant in the past two years.
4. Patients with pulmonary lymphangitic involvement that results in pulmonary dysfunction requiring active treatment, including the use of oxygen
5. Patients with active symptomatic brain metastases. Patients with central nervous system (CNS) metastases are considered eligible if they have had adequately treated brain metastases, ie, have completed treatment (tapered off steroids) at least four weeks before starting treatment with E7389. Patients who have no evidence that the metastases are symptomatic or actively growing (no evidence of midline shift on computed tomography scan or magnetic resonance imaging) may be enrolled without initiation of local therapy for the CNS metastases. In this case, a repeat scan must be performed within four weeks of the original scan to ensure that disease progression is not occurring. It is not the intention of this study to treat patients with active brain metastases.
6. Patients with meningeal carcinomatosis.
7. Patients who require therapeutic anti-coagulant therapy with warfarin or related compounds.
8. Women who are pregnant or breast-feeding. Women of childbearing potential with either a positive pregnancy test at Screening or no pregnancy test. Women of childbearing potential unless (1) surgically sterile or (2) using adequate measures of contraception in the opinion of the investigator (e.g., using 2 forms of contraception including a barrier method). Perimenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential.
9. Fertile men who are not willing to use contraception or fertile men with a female partner who is not willing to use contraception.
10. Patients with severe/uncontrolled intercurrent illness or infection.
11. Patients with significant cardiovascular impairment (history of congestive heart failure > New York Heart Association Grade II, unstable angina or myocardial infarction within the past six months, or serious cardiac arrhythmia).
12. Patients with organ allografts.
13. Patients who have a history of positive testing for HIV and/or have active hepatitis B or active hepatitis C at study entry.
14. Patients with pre-existing neuropathy > Grade 2.
15. Patients with a hypersensitivity to halichondrin B and/or to a halichondrin B chemical derivative.
16. Patients who participated in a prior E7389 clinical trial.
17. Patients with other significant disease or disorders that, in the investigator's opinion, would exclude the patient from the study.

For NSCLC patients at the MTD, the following additional exclusion criterion must be fulfilled:

1. Patients who have had a prior malignancy, other than carcinoma in situ of the cervix, or non-melanoma skin cancer, unless the prior malignancy was diagnosed and definitively treated ≥ five years previously with no subsequent evidence of recurrence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2006-10; Primary Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eisai US Medical Services, Study Director — Eisai Inc.
Locations (11):
- United States (4):
  - New Brunswick, New Jersey
  - Lake Success, New York
  - New York, New York
  - The Bronx, New York
- Austria (3):
  - Graz
  - Salzburg
  - Vienna
- India (4):
  - Vijayawada, Andhra Pradesh
  - Pune, Maharashtra
  - New Delhi, National Capital Territory of Delhi
  - Melur, Tamil Nadu

REFERENCES:
- [Derived] Goel S, Swami U, Kumar K, Dittrich C, Reyderman L, Jain M, Aisner J, Song J, Petrylak DP. A phase 1b, multicenter, open-label, dose-finding study of eribulin in combination with carboplatin in advanced solid tumors and non-small cell lung cancer. Cancer Chemother Pharmacol. 2019 Sep;84(3):567-578. doi: 10.1007/s00280-019-03877-4. Epub 2019 Jun 12. PMID 31190276

RESULTS

PARTICIPANT FLOW:
Groups:
- Eribulin Mesylate Dose Finding Plus Carboplatin AUC 5: Eribulin mesylate dose finding plus carboplatin AUC 5 in subjects with advanced solid tumors
- Eribulin Mesylate Dose Finding Plus Carboplatin AUC 6: Eribulin mesylate dose finding plus carboplatin AUC 6 in subjects with advanced solid tumors
- Eribulin Mesylate 1.1 mg/m^2 Plus Carboplatin AUC 6: Eribulin mesylate 1.1 mg/m2 plus carboplatin AUC 6 in subjects with non small cell lung cancer (NSCLC)
Period: Overall Study
Arm/Group | Eribulin Mesylate Dose Finding Plus Carboplatin AUC 5 | Eribulin Mesylate Dose Finding Plus Carboplatin AUC 6 | Eribulin Mesylate 1.1 mg/m^2 Plus Carboplatin AUC 6
Started | 43 | 9 | 12
Completed | 0 | 0 | 0
Not Completed | 43 | 9 | 12
Not completed — Adverse Event | 3 | 0 | 4
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 3
Not completed — Progressive Disease | 28 | 4 | 3
Not completed — Physician Decision | 3 | 0 | 1
Not completed — Clinical Progression | 9 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eribulin Mesylate Dose Finding Plus Carboplatin AUC 5 | Eribulin Mesylate Dose Finding Plus Carboplatin AUC 6 | Eribulin Mesylate 1.1 mg/m^2 Plus Carboplatin AUC 6 | Total
Number analyzed (Participants) | 43 | 9 | 12 | 64
Age Continuous [Mean (Standard Deviation); unit: years] | 59.2 (8.35) | 60.9 (8.08) | 64.4 (10.04) | 60.4 (8.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 5 | 1 | 28
  Male | 21 | 4 | 11 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 5 | 5
  Black or African American | 14 | 5 | 0 | 19
  White | 23 | 3 | 7 | 33
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 1 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Eribulin Mesylate of E7389 in Combination With Carboplatin in Subjects With Advanced Solid Tumors.
Description: MTD was established by summarizing the number and percent of subject with dose- limiting toxicities (DLTs) for the first cycle.
Time Frame: 21 days (first cycle)
Measure: Number; unit: mg/m^2
Arm/Group | Eribulin Mesylate Dose Finding Plus Carboplatin AUC 5 | Eribulin Mesylate Dose Finding Plus Carboplatin AUC 6 | Eribulin Mesylate 1.1 mg/m^2 Plus Carboplatin AUC 6
Number analyzed (Participants) | 43 | 9 | 12
mg/m^2 | 1.4 | 1.1 | 1.1

2. Secondary Outcome: Safety of Eribulin Mesylate in Combination With Carboplatin as Measured by the Number of Subjects With Treatment Emergent Adverse Events.
Description: Adverse events were considered treatment emergent if they started on or after the date of administration of the first dose of study drug, or if they were present prior to the administration of the first dose of study drug and increased in severity during the study.
Time Frame: Throughout the entire study
Population: Safety Evaluable Population
Measure: Number; unit: participants
Arm/Group | Eribulin Mesylate Dose Finding Plus Carboplatin AUC 5 | Eribulin Mesylate Dose Finding Plus Carboplatin AUC 6 | Eribulin Mesylate 1.1 mg/m^2 Plus Carboplatin AUC 6
Number analyzed (Participants) | 43 | 9 | 12
participants | 42 | 9 | 12

3. Secondary Outcome: Percent of Subjects With Best Overall Response as Measured by Response Evaluation Criteria in Solid Tumors (RECIST) Criteria.
Description: Objective response measured by Response Evaluation Criteria In Solid Tumors (RECIST) criteria and is Complete Response (disappearance of all target lesions) plus Partial Response (at least 30% decrease in sum of longest diameter [LD] of target lesions compared baseline sum of LD).
Time Frame: From start of eribulin treatment until disease progression or death
Population: Efficacy Evaluable Population
Measure: Number; unit: percentage of subjects
Arm/Group | Eribulin Mesylate Dose Finding Plus Carboplatin AUC 5 | Eribulin Mesylate Dose Finding Plus Carboplatin AUC 6 | Eribulin Mesylate 1.1 mg/m^2 Plus Carboplatin AUC 6
Number analyzed (Participants) | 43 | 9 | 11
percentage of subjects
  Best Overall Response Rate | 7 | 11.1 | 27.3
  Complete Response | 2.3 | 0 | 0
  Partial Response | 4.7 | 11.1 | 27.3
  Stable Disease | 48.8 | 33.3 | 36.4
  Progressive Disease | 32.6 | 22.2 | 9.1
  Not Evaluable | 11.6 | 33.3 | 27.3

ADVERSE EVENTS:
Arm/Group | Eribulin Mesylate Dose Finding Plus Carboplatin AUC 5 | Eribulin Mesylate Dose Finding Plus Carboplatin AUC 6 | Eribulin Mesylate 1.1 mg/m^2 Plus Carboplatin AUC 6
Serious Adverse Events (participants affected / at risk) | 18/43 | 5/9 | 8/12
Other Adverse Events (participants affected / at risk) | 42/43 | 9/9 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eribulin Mesylate Dose Finding Plus Carboplatin AUC 5 (N=43) | Eribulin Mesylate Dose Finding Plus Carboplatin AUC 6 (N=9) | Eribulin Mesylate 1.1 mg/m^2 Plus Carboplatin AUC 6 (N=12)
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 3
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 3
Cardiac Failure (Cardiac disorders) | 0 | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1
Infection (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 2
Radius Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Oral Intake Reduced (Metabolism and nutrition disorders) | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Malignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebral Hemorrhage (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Sensorimotor Disorder (Nervous system disorders) | 1 | 0 | 0
Spinal Cord Compression (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Syringomyelia (Nervous system disorders) | 1 | 0 | 0
Cerebral Ischemia (Nervous system disorders) | 0 | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 1 | 0 | 1
Renal Vein Thrombosis (Renal and urinary disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 2 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eribulin Mesylate Dose Finding Plus Carboplatin AUC 5 (N=43) | Eribulin Mesylate Dose Finding Plus Carboplatin AUC 6 (N=9) | Eribulin Mesylate 1.1 mg/m^2 Plus Carboplatin AUC 6 (N=12)
Anemia (Ear and labyrinth disorders) | 15 | 2 | 7
Leukopenia (Blood and lymphatic system disorders) | 4 | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 22 | 6 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 16 | 2 | 8
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 4
Cardiac Failure (Cardiac disorders) | 0 | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 0 | 0 | 1
Sinus Tachycardia (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Conjunctival Hyperaemia (Eye disorders) | 0 | 0 | 1
Abdominal Distention (Gastrointestinal disorders) | 3 | 7 | 2
Abdominal Pain (Gastrointestinal disorders) | 9 | 1 | 1
Constipation (Gastrointestinal disorders) | 10 | 4 | 4
Diarrhea (General disorders) | 11 | 1 | 4
Nausea (Gastrointestinal disorders) | 17 | 4 | 3
Vomiting (Gastrointestinal disorders) | 10 | 5 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 2 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1
Frequent Bowel Movements (Gastrointestinal disorders) | 0 | 0 | 1
GI Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 1
Melena (Gastrointestinal disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Tooth Loss (Gastrointestinal disorders) | 0 | 0 | 1
Gingival Pain (Gastrointestinal disorders) | 0 | 1 | 0
Hemorrhoidal Hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 23 | 7 | 8
Performance Status Decreased (Hepatobiliary disorders) | 6 | 2 | 0
Catheter Site Pain (General disorders) | 0 | 1 | 0
Gait Disturbance (General disorders) | 0 | 1 | 0
Edema Peripheral (General disorders) | 0 | 1 | 2
Asthenia (General disorders) | 0 | 1 | 1
Axillary Pain (General disorders) | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 1
Extravasation (Hepatobiliary disorders) | 0 | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 5
Urinary Tract Infection (Infections and infestations) | 3 | 1 | 0
Infusion Site Infection (Infections and infestations) | 0 | 1 | 0
Localised Infection (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1
Candidiasis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 1
Oral Candidiasis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Nervous system disorders) | 0 | 0 | 2
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femural Neck Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood Lactate Dehydrogenase Increased (Metabolism and nutrition disorders) | 3 | 0 | 0
Weight Decreased (Investigations) | 6 | 1 | 3
Alanine Aminotransferase Increased (Investigations) | 0 | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 1 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 1 | 0
Breath Sounds Abnormal (Investigations) | 0 | 2 | 0
Neutrophil Count Decreased (Investigations) | 0 | 1 | 0
Hemoglobin Decreased (Investigations) | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 10 | 5 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 0 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 3 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1
Oral Intake Reduced (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 4 | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1
Myalgia (Nervous system disorders) | 4 | 0 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 5 | 1 | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Dizziness (Nervous system disorders) | 6 | 0 | 2
Dysgeusia (Nervous system disorders) | 3 | 0 | 1
Headache (Nervous system disorders) | 6 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 3 | 1 | 0
Neuropathy Peripheral (Nervous system disorders) | 4 | 0 | 2
Ageusia (Nervous system disorders) | 0 | 1 | 0
Amnesia (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Areflexia (Nervous system disorders) | 0 | 1 | 0
Hypogeusia (Nervous system disorders) | 0 | 1 | 0
Insomnia (Nervous system disorders) | 0 | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Restless Leg Syndrome (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Cerebral Ischemia (Nervous system disorders) | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 1
Neuropathy (Nervous system disorders) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 3 | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 5
Dyspnea (Skin and subcutaneous tissue disorders) | 7 | 3 | 5
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dysphonia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dyspnea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 3 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 0 | 0
Facial Wasting (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pain in Skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash Poplar (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 2 | 1
Hematoma (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 2
Flushing (Vascular disorders) | 0 | 0 | 1
Phlebitis (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No